CLINICAL TRIAL: NCT06559007
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Single Dose HRS-5041 in Healthy Caucasian Male Participants
Brief Title: Phase 1 Study to Evaluate PK, Safety, and Tolerability of HRS-5041 in Healthy Caucasian Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5041-102
Record Dates: First submitted 2024-08-02; First posted 2024-08-19 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Administration, Oral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: HRS-5041 dose level 1 (Experimental): Sing dose level 1
  Interventions: Drug: HRS-5041 dose level 1
- Experimental: HRS-5041 dose level 2 (Experimental): Sing dose level 2
  Interventions: Drug: HRS-5041 dose level 2

INTERVENTIONS:
Drug: HRS-5041 dose level 1 — Single dose of HRS-5041 orally administered
  Other Names: HRS-5041 (single dose, oral administration, dose level 1)
  Arms: Experimental: HRS-5041 dose level 1
Drug: HRS-5041 dose level 2 — Single dose of HRS-5041 orally administered
  Other Names: HRS-5041 (single dose, oral administration, dose level 2)
  Arms: Experimental: HRS-5041 dose level 2

SUMMARY:
This is a phase 1, open-label, randomized study. The objective of this study is to evaluate the PK, safety and tolerability of orally administered single-dose HRS-5041 in healthy Caucasian male participants.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the PK, safety and tolerability of orally administered single-dose HRS-5041 in healthy Caucasian male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian participants;
2. Ability to understand the trial procedures and possible adverse events, voluntarily participate in the trial,
3. Male aged between 18 to 55 years of age (inclusive) at the date of signed consent form.
4. Total body weight ≥ 50.0 kg, body mass index (BMI) between 19.0 and 32.0 kg/m2 (inclusive) at screening.

Exclusion Criteria:

1. History of receiving any androgen receptor (AR) degraders.
2. History or evidence of clinically significant
3. History of severe abnormal gastric emptying, severe gastrointestinal (GI) disease, or participants who had GI surgeries (except GI polypectomy).
4. Severe infections, injuries, or major surgeries as determined by the investigator within 6 months
5. Any other circumstances (e.g., not suitable for venous access) or laboratory abnormality that, in the investigator's judgment, may increase the risk to the participant, or be associated with the participant's participation in and completion of the study or could preclude the evaluation of the participant's response.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
PK profile (Cmax) of HRS-5041 after a single oral (PO) administration: | Day 10
  Parameters: Cmax
PK profile (AUC0-t) of HRS-5041 after a single oral (PO) administration: | Day 10
  Parameter: AUC0-t
PK profile (AUC0-inf) of HRS-5041 after a single oral (PO) administration: | Day 10
  Parameter:AUC0-inf
PK profile (Tmax) of HRS-5041 after a single oral (PO) administration: | Day 10
  Parameter: Tmax
PK profile ( t1/2) of HRS-5041 after a single oral (PO) administration: | Day 10
  Parameter: t1/2
PK profile (CL/F) of HRS-5041 after a single oral (PO) administration: | Day 10
  Parameter: CL/F
PK profile (Vz/F) of HRS-5041 after a single oral (PO) administration: | Day 10
  Parameter: Vz/F

SECONDARY OUTCOMES:
Safety and tolerability - number and severity of adverse events | Day 10
  Incidence and severity of AE
Safety and tolerability - Blood pressure | Day 10
  Incidence of Adverse Events and Abnormalities as assessed by blood pressure (systolic and diastolic pressure)
Safety and tolerability - Body temperature | Day 10
  Incidence of Adverse Events and Abnormalities as assessed by body temperature
Safety and tolerability - Physical examination | Day 10
  Incidence of Adverse Events and Abnormalities as Assessed by Physical Examination
Safety and tolerability - Laboratory tests | Day 10
  Number of abnormalities assessed based on safety bloods and urine test
Safety and tolerability - ECG | Day 10
  heart rate, PR interval, QT interval, corrected QT (QTcF using Fridericia's formula) interval, and QRS

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Melbourne, Melbourne, Victoria, Australia